CLINICAL TRIAL: NCT05987904
Title: MDR - Feasibility Study for Instant Cardiac Diagnostic and Post-operative Risk
Brief Title: Feasibility Study for Instant Cardiac Diagnostic and Post-operative Risk Assessment with the LynxPatch Device
Acronym: LP-I-CARDIAG
Status: Completed | Type: Observational
Sponsor: Lynx Health Science GmbH (Industry)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MDR LP-I-CARDIAG
Record Dates: First submitted 2023-07-28; First posted 2023-08-14 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases
Keywords: Cardiac Diagnosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Cardiologic Group: This group includes patients who are scheduled for echocardiography.
  Interventions: Device: LynxPatch
- Group 2: Surgery Group: This group includes patients that are scheduled for non-cardiac surgery.
  Interventions: Device: LynxPatch

INTERVENTIONS:
Device: LynxPatch — Measurements with the LynxPatch device are conducted.

SUMMARY:
In this clinical study the investigators will evaluate if it is feasible to pre-operatively identify low-risk patients, and to identify patients with cardiac pathologies with the LynxPatch.

DETAILED DESCRIPTION:
The LynxPatch is a non-invasive, wireless device for cardiac diagnosis. The aim of this study is to compare the LynxPatch predictions with the echocardiographic diagnoses of cardiac pathologies and to evaluate its perioperative risk predictions in non-cardiac surgeries. The study population includes 1100 patients that scheduled for an echocardiographic assessment or for a non-cardiac surgery. The LynxPatch measurement procedure has a duration of about 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent, i.e., the subject must be able to understand and sign the Patient Information and Consent Form.
* Group 1: Patients that have an indication for an echocardiographic assessment.
* Group 2: Patients that are scheduled for a non-cardiac surgery

Exclusion Criteria:

* Subjects has implanted cardioverter defibrillator
* Subject is pregnant
* Subject is breastfeeding
* Subject has compromised skin in the location where the LynxPatch is intended to be positioned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, all patients will be consecutively recruited that are either scheduled for an echocardiographic examination or that will be subjected to a non-cardiac surgical procedure according to their respective standard procedure.
Sampling Method: Non-Probability Sample
Enrollment: 1097 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Level of agreement between the LynxPatch device and echocardiography in detecting a cardiac pathology. | 30 minutes per individual
  Comparison of the detection of the presence of a cardiac pathology by the LynxPatch device and by echocardiography-based expert diagnosis.

SECONDARY OUTCOMES:
Accuracy of the LynxPatch device predictions of an adverse perioperative outcome | 30 days per individual
  Comparison of the LynxPatch device predictions of an adverse perioperative outcome with actually occuring adverse perioperative outcome.
Usability of the LynxPatch device | 30 minutes per individual
  Evaluation of aspects of the LynxPatch device's usability by interviewing study participants using a questionnaire.
Rate of LynxPatch-related safety incidents | 30 minutes per individual
  Assessment of safety-related aspects with the LynxPatch device. Relevant incidents include Adverse Device Effects, Serious Adverse Device Effects and Device Defficiencies.

CONTACTS AND LOCATIONS:
Overall Officials: Aydan Ewers, Dr. med., Principal Investigator — BG Universitätsklinikum Bergmannsheil
Locations (1):
- Med. Klinik II - Kardiologie und Angiologie, Bochum, Germany

IPD SHARING:
Plan to Share IPD: No